CLINICAL TRIAL: NCT04192500
Title: A Phase 2a, Single Center, Randomized, Double-blind, Controlled Study to Evaluate the Immunogenicity and the Safety of One Dose of OVX836 Influenza Vaccine at Two Dose Levels (90 µg and 180 μg), in Comparison to Influvac TetraTM, Quadrivalent Seasonal Influenza Sub-unit Vaccine, After Intramuscular Administration in Healthy Subjects Aged 18-65 Years
Brief Title: Safety and Immune Response of One Dose of OVX836 at Two Dose Levels, in Comparison to Influvac TetraTM, After Intramuscular Administration in Healthy Subjects Aged 18-65 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Osivax (Industry)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OVX836-002
Record Dates: First submitted 2019-12-03; First posted 2019-12-10 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Randomized assignment to experimental vaccine (2 dosage levels or active control (commercial influenza vaccine) in a 1:1:1 ratio.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- OVX836 - 90µg dose (Experimental): Adjuvant-free recombinant influenza candidate vaccine based on the Nucleoprotein (NP) of the influenza virus. One single administration intramuscularly of a 90µg dose on Day 1.
  Interventions: Biological: OVX836
- OVX836 - 180µg dose (Experimental): Adjuvant-free recombinant influenza candidate vaccine based on the Nucleoprotein (NP) of the influenza virus. One single administration intramuscularly of a 180µg dose on Day 1.
  Interventions: Biological: OVX836
- Quadrivalent seasonal influenza vaccine (Influvac TetraTM) (Active Comparator): Licensed quadrivalent seasonal influenza subunit vaccine for season 2019-2020. One full dose to be administered at Day 1
  Interventions: Biological: Quadrivalent seasonal influenza vaccine (Influvac TetraTM)

INTERVENTIONS:
Biological: OVX836 — One single administration intramuscularly at Day 1.
  Arms: OVX836 - 180µg dose; OVX836 - 90µg dose
Biological: Quadrivalent seasonal influenza vaccine (Influvac TetraTM) — One single administration intramuscularly at Day 1.
  Arms: Quadrivalent seasonal influenza vaccine (Influvac TetraTM)

SUMMARY:
This Phase 2a clinical study is designed to evaluate the immunogenicity and the safety of one dose of OVX836 influenza vaccine administered IM, confirm the dose level and regimen, and expand immunogenicity and safety data to adults through age 65.

DETAILED DESCRIPTION:
This is a Phase 2a, randomised, double-blind study in 300 adults to compare the safety and immunogenicity of OVX836 to QIV (Influvac TetraTM). One dose of OVX836 at two dose levels will be administered intramuscularly, in comparison to Influvac TetraTM, quadrivalent seasonal influenza sub-unit vaccine in healthy subjects aged 18-65 years.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Healthy male or female subjects, as determined by medical history and medical examination.
3. Between the ages of 18 and 65 years, inclusive.
4. Reliable and willing to make themselves available for the duration of the study, and willing and able to follow study procedures.

Exclusion Criteria:

1. Subject with a body mass index (BMI) ≥35 kg/m² on the day of vaccination.
2. Previous influenza vaccination within 6 months before the day of vaccination, or planned to receive during the study duration.
3. Any known or suspected immunodeficient conditions.
4. Past or current history of significant autoimmune diseases, as judged by the Investigator.
5. Current history of significant uncontrolled medical illness such as diabetes, hypertension, heart, renal or hepatic diseases, as judged by the Investigator.
6. Female subjects: pregnant, breast-feeding or of childbearing potential without appropriate contraceptive methods in place for 2 months before enrolment, or with positive pregnancy test on the day of vaccination. Appropriate contraceptive methods are defined by the Clinical Trial Facilitation Group [CTFG] as follow: "Contraceptive methods that can achieve a failure rate of less than 1% per year when used consistently and correctly are considered as highly effective birth control methods. Such methods include: combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable intrauterine device, intrauterine hormone-releasing system), bilateral tubal occlusion, vasectomized partner and/or sexual abstinence (refraining from heterosexual intercourse)."
7. Having received another vaccination within 3 months prior to the day of study vaccination for live attenuated vaccines, or within 1 month prior to the day of study vaccination for inactivated vaccines.
8. Planning to receive other vaccines during the first 28 days following the study vaccine administration.
9. Administration of any investigational or non-registered drug or vaccine within 3 months prior to the administration of study vaccines, or planned administration of any such product during the whole study period.
10. History of receiving blood, blood components or immunoglobulins within 3 months prior to the day of vaccination, or planned to receive such product during the whole study period.
11. Presence of an acute febrile illness on the day of vaccination (oral temperature >38.0°C, temporary exclusion criterion).
12. Past or current history of any progressive or severe neurological disorder, seizure disorder or Guillain-Barré syndrome.
13. Behavioral or cognitive impairment, or psychiatric disease that, in the opinion of the Investigator, may interfere with the subject's ability to participate in the study.
14. Past (stopped less than 6 months before enrolment) or current history of alcohol or drug abuse, or current smoking habit above 10 cigarettes per day.
15. Treatment that can affect immune response such as systemic or high dose inhaled corticosteroids (>800 μg/day beclomethasone or equivalent; occasional inhaled corticosteroids for asthma therapy are allowed), radiation treatment, cytotoxic drugs, or current or recent (within 30 days before study entry) chronic or prolonged (>10 days) use of systemic non-steroidal anti-inflammatory drugs, interferon, immunomodulators, allergy shots, as judged by the Investigator.
16. Subjects with known or suspected anemia.
17. Recent blood or platelets donation (less than 3 months before enrolment). History of plasma donation is authorized.
18. History of severe allergic reactions and/or anaphylaxis, or serious adverse reactions to vaccines or allergy to kanamycin, or to any component that may be present in the comparator vaccine, as traces such as eggs (ovalbumin, chicken proteins), formaldehyde, cetyltrimethylammonium bromide, polysorbate 80, or gentamicin.
19. Any contraindication to intramuscular administration, as judged by the Investigator.
20. Individuals with history of any illness that, in the opinion of the Investigator, might interfere with the results of the study or pose additional risk to the subjects due to participation in the study.
21. Technical difficulties in the use of an e-diary.
22. Sponsor employees or Investigator site personnel directly affiliated with this study, and their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2020-09-07 (Actual); Study Completion 2020-09-07 (Actual)

PRIMARY OUTCOMES:
NP-specific IFNγ T-cell increase measured by ELISPOT at Day 8 versus pre-injection baseline (Day 1) in the pooled age strata | at Day 8 versus pre-injection baseline (Day 1)

SECONDARY OUTCOMES:
Proportion of subjects reporting solicited local (Injection site redness, Injection site swelling, Injection site pain) and systemic symptoms (Fatigue, Headache, Arthralgia, Malaise, Myalgia, Fever) using an electronic Diary | during 7 days after vaccine administration
Proportion of subjects reporting unsolicited Adverse Events | during 28 days after vaccine administration
Proportion of subjects with Influenza-Like-Illness cases associated with laboratory-confirmed influenza | during the whole study duration, 180 days
Severity scores of Influenza-Like-Illness cases (as per Flu-PRO® questionnaire) | during the whole study duration, 180 days
Proportion of subjects reporting Serious Adverse Events | during the whole study duration, 180 days
NP-specific IFNγ T-cell activity measured by ELISPOT in the pooled age strata and by age stratum (18-49 years; 50-65 years) | at Day 8, Day 29 and Day 180 versus pre-injection baseline (Day 1)
NP T-cell phenotype and functionality by flow cytometry in the pooled age strata and by age stratum (18-49 years; 50-65 years) | at pre-injection baseline (Day 1), Day 8, Day 29 and Day 180
Anti-NP Immunoglobulin G (IgG) titers by ELISA at each time point in the pooled age strata and by age stratum (18-49 years; 50-65 years) | at pre-injection baseline (Day 1), Day 8, Day 29 and Day 180

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Leroux-Roels, MD, PhD, Principal Investigator — Centre for Vaccinology (CEVAC), Ghent University Hospital
Locations (1):
- Centre for Vaccinology (CEVAC), Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leroux-Roels I, Waerlop G, Tourneur J, De Boever F, Maes C, Bruhwyler J, Guyon-Gellin D, Moris P, Del Campo J, Willems P, Leroux-Roels G, Le Vert A, Nicolas F. Randomized, Double-Blind, Reference-Controlled, Phase 2a Study Evaluating the Immunogenicity and Safety of OVX836, A Nucleoprotein-Based Influenza Vaccine. Front Immunol. 2022 Apr 7;13:852904. doi: 10.3389/fimmu.2022.852904. eCollection 2022. PMID 35464450
- See also: Randomized, Double-Blind, Reference-Controlled, Phase 2a Study Evaluating the Immunogenicity and Safety of OVX836, A Nucleoprotein-Based Influenza Vaccine — https://pubmed.ncbi.nlm.nih.gov/35464450/